CLINICAL TRIAL: NCT06503978
Title: Dosing Study of Microbiota Transplant Therapy for Children With Autism Spectrum Disorder (ASD) Who Have Gastrointestinal Disorders
Brief Title: Microbiota Transplant Therapy for Children With Both Autism Spectrum Disorder and Gastrointestinal Disorders
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gut-Brain-Axis Therapeutics Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WCG IRB #20242031
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder; Gastro-Intestinal Disorder; Constipation; Diarrhea
Keywords: fecal transplant; fecal microbiota transplant
MeSH Terms: conditions — Autism Spectrum Disorder; Digestive System Diseases; Constipation; Diarrhea | interventions — Vancomycin; polyethylene glycol 3350; Antacids

STUDY DESIGN:
Intervention Model Description: Part 1: Randomized, Double-Blinded, Placebo-Controlled with 2 Treatment groups and 2 Placebo Groups (15 weeks)
  Part 2: Open-Label Observation and Cross-over or Treatment Part 3: Follow Up (Group B Only)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, Investigators and outcome assessors were all blinded. Only the Pharmacist distributing the medication knew the randomization code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A: Treatment (Dose 1) (Experimental): Part 1: Blinded Treatment (15 weeks)
  Vancomycin, Miralax, Antacid, MTP-101P
  Interventions: Combination Product: MTP-101P; Combination Product: Vancomycin; Combination Product: Miralax; Combination Product: Antacid
- Group B: Treatment (Dose 2) (Experimental): Part 1: Blinded Treatment (15 weeks)
  Vancomycin, Miralax, Antacid, MTP-101P
  Interventions: Combination Product: MTP-101P; Combination Product: Vancomycin; Combination Product: Miralax; Combination Product: Antacid
- Group C: Placebo (Placebo Comparator): Part 1: Blinded Placebo (15 weeks)
  Placebo Vancomycin, Real Miralax, Real Antacid, Placebo MTP-101P
  Interventions: Combination Product: Miralax; Combination Product: Placebo MTP-101P; Combination Product: Placebo Vancomycin
- Group D: Placebo (Placebo Comparator): Part 1: Blinded Placebo (15 weeks)
  Placebo Vancomycin, Real Miralax, Real Antacid, Placebo MTP-101P
  Interventions: Combination Product: Miralax; Combination Product: Placebo MTP-101P; Combination Product: Placebo Vancomycin

INTERVENTIONS:
Combination Product: MTP-101P — MTP-101P is comprised of standardized dose of total fecal microbiota purified from the stool of healthy donors. Donors are carefully screened via health status questionnaires, physical examinations, reviews of comprehensive medical history, clinical laboratory evaluations, serologic and genomic tests for infectious diseases and metabolic health, and stool-related pathogen testing. The material from the donors is purified to remove the majority of non-bacterial material, washed, lyophilized, and provided to the patient in a sachet contained within a mixing bottle.
  Arms: Group A: Treatment (Dose 1); Group B: Treatment (Dose 2)
Combination Product: Vancomycin — Oral vancomycin is an antibiotic used for treating C. difficile-associated diarrhea and staphylococcal-induced enterocolitis.
  Duration: 14 Days
  Arms: Group A: Treatment (Dose 1); Group B: Treatment (Dose 2)
Combination Product: Miralax — Miralax is a common over-the-counter laxative and bowel cleanse
Combination Product: Antacid — The antacid will be aluminum/magnesium hydroxide, 1x/day, 5 minutes before the MTP-101P. Each 5 ml consists of Aluminum Hydroxide - 200 mg, Magnesium Hydroxide - 200 mg, and Simethicone - 20 mg. If some participants cannot tolerate the aluminum/magnesium hydroxide, we will allow calcium carbonate alternatives equivalent in acid neutralizing capacity.
  Duration: 12 weeks
  Arms: Group A: Treatment (Dose 1); Group B: Treatment (Dose 2)
Combination Product: Placebo MTP-101P — The same packaging will be used as for MTP-101P, but the sachets will contain a freeze-dried mixture of normal saline containing 10% Trehalose.
  Duration: 12 weeks
  Arms: Group C: Placebo; Group D: Placebo
Combination Product: Placebo Vancomycin — Same packaging and liquid carrier and flavoring used as for the oral vancomycin, but no vancomycin.
  Duration: 14 days
  Arms: Group C: Placebo; Group D: Placebo

SUMMARY:
The investigators propose to investigate Microbiota Transfer Therapy (MTT) for treating patients with Autism-spectrum disorder with Gastrointestinal disorders (constipation, diarrhea, and/or abdominal pain). MTT involves a combination of 14 days of oral vancomycin (an antibiotic to kill pathogenic bacteria), followed by 1 day of bowel cleanse using Miralax, followed by 5 days of high dose MTP-101P with an antacid, followed by 12 weeks of a lower maintenance dose of MTP-101P with an antacid.

DETAILED DESCRIPTION:
For children 4 to less than <18 years old with Autism-spectrum disorder with Gastrointestinal disorders (constipation, diarrhea, and/or abdominal pain). This will be a Phase 2 randomized controlled trial to compare two dosing strategies for microbiota transplant vs. placebo.

Participants will be randomly assigned to Group A, B, C or D

Part 1: Placebo-Controlled Treatment (15 Weeks) The trial will begin with a randomized, double-blind, placebo-controlled trial which will include a 14-day treatment with oral vancomycin (or placebo), then 1 day of Miralax to cleanse the bowel of vancomycin and bacteria/feces (all participants, since its bowel-emptying effect cannot be blinded), followed by 5 days of initial high dose of MTP-101P taken daily 5 minutes after antacid, and then 12 weeks of a lower maintenance dose of MTP-101P taken daily 5 minutes after an antacid.

Group A: Real Treatment. Dose 1 Group B: Real Treatment. Dose 2 Group C: Placebo vancomycin, real Miralax, placebo MTP-101P, real antacid. Group D: Placebo vancomycin, real Miralax, placebo MTP-101P, real antacid.

Part 2: Open-Label Observation and Cross-Over (12 weeks)

Group A: Observation over the next 12 weeks (no additional treatment). Group B: Observation over the next 12 weeks (no additional treatment). Group A and B completes study at end of part 2.

Group C will receive the same dosage group A received in part 1 (Dose 1). This includes 14 days of vancomycin, Miralax, and an initial high dose of MTP-101P for 5 days taken daily 5 minutes after an antacid, and then a lower dose of MTP-101P for 12 weeks taken daily 5 minutes after antacid.

Group D will receive the same dosage group B received in part 1 (Dose 2). This includes 14 days of vancomycin, Miralax, and an initial high dose of MTP-101P for 5 days taken daily 5 minutes after an antacid, and then a lower dose of MTP-101P for 12 weeks taken daily 5 minutes after antacid.

Part 3: Follow Up Group C and D. There will be a follow-up evaluation 15 weeks post-treatment after the end of Part 2, to assess long-term efficacy and possible adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Child aged 4 to < 18 years. This is 1 year younger than our previous study of MTT for children with ASD (IND 19048, protocol 2), because there were minimal adverse effects in that study, and earlier intervention may be more beneficial.
2. Diagnosis of autism per the Childhood Autism Rating Scale 2 (CARS-2) and either the Autism Diagnostic Interview-Revised (ADI-R) or the Autism Diagnostic Observation Schedule 2 (ADOS 2).
3. GI disorder as defined below that has lasted for at least 1 year.
4. No changes in medications, supplements, diet, therapies, or education in the 2 months prior to starting treatment, and no intention to change them during the clinical trial.
5. General good physical health aside from gastrointestinal problems.
6. At least two previous trials of "standard of care" GI treatments that did not alleviate GI symptoms (constipation, diarrhea, bloating, gas, reflux, and/or abdominal pain). Standard of care treatments include laxatives, stool softeners, enemas, suppositories, or similar medications.

Exclusion Criteria:

1. Antibiotics in 3 months prior to treatment (does not apply to topical antibiotics).
2. Probiotics in 2 months prior to treatment, or fecal transplant in previous 12 months. Foods naturally containing probiotics such as yogurt are allowed.
3. Single-gene disorder (Fragile X, etc.).
4. Major brain malformation.
5. Tube feeding.
6. Current severe gastrointestinal problems that require immediate treatment (life-threatening).
7. Severely underweight/malnourished (per physician clinical judgement).
8. Unstable, poor health; seizure disorder that is not responsive to treatment or not on stable management or complex type; or other health conditions that would significantly increase their risk of adverse effects (per physician clinical judgement) including active malignancy or infection.
9. Recent or scheduled surgeries.
10. Ulcerative Colitis, Crohn's Disease, diagnosed Celiac Disease, Eosinophilic Gastroenteritis, or similar conditions.
11. Current participation in other clinical trials.
12. Females who are pregnant or who are at risk of pregnancy and sexually active with a male partner without effective birth control. We will conduct a pregnancy test on all female participants 12 years and older as part of the screening and at each clinical visit.

    a. Males who are sexually active with a female partner without highly effective birth control (IUD or birth control hormones).
13. Allergy or intolerance to the study medications: vancomycin, Miralax, milk powder with soy and chocolate flavoring (which are included in MTP-101P), or the antacid. People with a known allergy or intolerance to milk, soy, or chocolate will be excluded from the study and will not participate in the tolerance test.
14. Clinically significant abnormalities at baseline on blood safety tests: Comprehensive Metabolic Panel and Complete Blood Count with Differential. If there is a clinically significant result, a second test may be used to confirm that result at the physician's discretion.
15. Psychotropic medication daily use - Current or within 2 months prior to treatment - which are known to interfere in gastrointestinal function.
16. Evidence of significant impairment of immune system, or taking medications that can compromise the immune system, and thus increase risk if exposed to multiple-drug resistant bacteria.
17. Substantially decreased kidney function, as evidenced by estimated glomerular filtration rate of <60 mL/min/1.73 m2. This is not normally reported for children on standard laboratory metabolic panels, so in those cases we will use the National Kidney Foundations Pediatric GFR Calculator to calculate the pediatric GFR based on age/height, the BUN and serum creatinine from our standard CMP (National Kidney Foundation Inc., n.d.). This calculator uses the Creatinine-based "Bedside Schwartz" equation (2009) that seems to be the most commonly used calculation for this purpose.
18. Participants who are breastfeeding.

The rational for exclusions 1-2 is that they interfere with gut flora. The rationale for exclusions 3-4 is that those individuals are probably less likely to respond to the proposed treatment.

The rationale for exclusions 5-9 is that those individuals are at higher risk of safety problems with MTT.

The rational for exclusion 10 is that inclusion of people with these GI conditions would complicate analysis of the study results.

The rational for exclusion 11 is that participation in other trials would interfere with the results of this one.

The rationale for exclusion 12 is to avoid risk to fetuses. The rationale for exclusion 13 is to avoid known allergic reactions to study medications.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-07-17 (Estimated); Study Completion 2026-08-17 (Estimated)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale (CARS-2) | Baseline (0-30 days prior to treatment) vs End of Treatment (Day 104)
  A 15-item scale that can be used to both diagnose autism and ASD and to assess the overall severity of symptoms
Daily Stool Record (DSR) | Screening (0-120 days prior to Baseline) vs Baseline (0-30 days prior to treatment) vs End of Treatment (Day 104)
  Participants will report the number of abnormal events during a 14 day period. An event includes no bowel movement during 1 day, unusually hard stool (Bristol Stool Form type 1-2), unusually soft stool (Bristol Stool Form type 6-7), four or more bowel movements in 1 day, abdominal pain, or use of GI medication. The units are number of events regardless of type of event.

SECONDARY OUTCOMES:
Gastrointestinal Symptom Rating Scale (GSRS) | Baseline (0-30 days prior to treatment) VS Day 14, 28,56,84 and 104
  An assessment of GI symptoms based on 15 questions, which are then scored in five domains (abdominal pain, reflux, indigestion, diarrhea, and constipation). Symptoms are rated on a 7-point Likert scale including no discomfort at all (1), slight discomfort (2), mild discomfort (3), moderate discomfort (4), moderately severe discomfort (5), severe discomfort (6), and very severe discomfort (7).
Clinical Global Impression - Gastrointestinal (CGI-GI) | Baseline (0-30 days prior to treatment) VS End of Treatment (Day 104)
  This assessment is conducted by the study physician and assess the severity of GI symptoms on a 7-point scale. The severity scale rates the severity of the patient's illness including normal, not at all ill (1), borderline mentally ill (2), mildly ill (3), moderately ill (4), markedly ill (5), severely ill (6), among the most extremely ill patients (7).
Clinical Global Impression - Autism (CGI-A) | Baseline (0-30 days prior to treatment) VS End of Treatment (Day 104)
  This assessment is conducted by the study physician and assess the severity of Autism Symptoms on a 7-point scale. The severity scale rates the severity of the patient's illness including normal, not at all ill (1), borderline mentally ill (2), mildly ill (3), moderately ill (4), markedly ill (5), severely ill (6), among the most extremely ill patients (7).
National Survey on treatment Effectiveness for Autism (NSTEA) | End of Treatment (Day 104)
  Assess the effectiveness of MTT on overall benefit (no benefit (0)/slight benefit(1)/moderate benefit (2)/good benefit (3)/great benefit (4)).
Social Responsiveness Scale (SRS 2) | Baseline (0-30 days prior to treatment) VS End of Treatment (Day 104)
  65-item scale that assesses social impairments, a core issue in autism, including social awareness, social information processing, capacity for reciprocal social communication, social anxiety/avoidance, and autistic preoccupations and traits.
Aberrant Behaviour Checklist (ABC-2) | Baseline (0-30 days prior to treatment) VS End of Treatment (Day 104)
  assesses problem behaviors in five areas common in individuals with ASD, including irritability, social withdrawal, stereotypic behavior, hyperactivity/noncompliance, and inappropriate speech.
CAAAS (subscale on GI symptoms) | Baseline (0-30 days prior to treatment) VS Day 14, 28,56,84 and 104
  This tool assesses both core ASD symptoms and a comprehensive list of common co-occurring symptoms in ASD, including gastrointestinal, behavioral, mental health, and physical health symptoms.
  9-point severity scale from "none" to "major". There is also a "change"
Comprehensive Assessment of Autism and Associated Symptoms (CAAAS) | Baseline (0-30 days prior to treatment) VS Day 14, 28,56,84 and 104
  This tool assesses both core ASD symptoms and a comprehensive list of common co-occurring symptoms in ASD, including gastrointestinal, behavioral, mental health, and physical health symptoms.
  9-point severity scale from "none" to "major". There is also a "change"
Vineland Adaptive Behavior Scale -Third Edition (Vineland 3) | Baseline (0-30 days prior to treatment) VS End of Treatment (Day 104)
  Comprehensive form consisting of 381 items covering three domains (Communication, Daily Living Skills, and Socialization) and the Maladaptive Behavior subscale (44 items).

CONTACTS AND LOCATIONS:
Locations (1):
- Autism/Asperger's Research Group at Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No